CLINICAL TRIAL: NCT06003972
Title: Asses the Anti-inflammatory Effects of Short Term Copaxone Therapy on Patients the Acute Decompensated Heart Failure
Acronym: Copaxone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, RABEA ASLEH, Professor, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 093418-HMO-CTIL
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Acute Decompensated Heart Failure; Cytokine Storm; Inflammatory Response; Heart Failure
MeSH Terms: conditions — Cytokine Release Syndrome; Heart Failure | interventions — Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): This arm serves as the control arm, patients allocated receive guideline directed medical therapy only
  Interventions: Drug: guideline directed medical therapy (GDMT)
- Copaxone arm (Experimental): Patients receive guideline directed medical therapy with an add-on GA therapy for 14 days
  Interventions: Drug: Copaxone

INTERVENTIONS:
Drug: Copaxone — Paptients allocated to this arm receive 20 mg GA given s.c daily for a total of 14 days
  Other Names: Glatiramer Acetate
  Arms: Copaxone arm
Drug: guideline directed medical therapy (GDMT) — GDMT for heart failure according to the AHA guidelines.
  Arms: Control

SUMMARY:
Assess the anti-inflammatory effects of short-term Copaxone therapy on patients with acute decompensated heart failure.

Trial Design

* An open-label, randomized, prospective trial of patients hospitalized due to acute decompensation of heart failure with reduced ejection fraction.
* Patients will be enrolled within 24 hours from hospital admission.
* Randomization and intervention will begin within 24 hours of enrollment (and at least 24 hours after admission).
* Patients will be randomized in a 1:1 ratio either to receive guideline directed medical therapy (GDMT) or GDMT plus Copaxone.
* Patients assigned to intervention group will receive daily SC Copaxone 20 mg for 14 days.
* Patients will be assessed during 4 time points(screening/randomization, visit 3 day, visit 14 day, visit 30 day) as elaborated in article "monitoring".
* Changes in inflammatory cytokines will be compared between control and intervention group throughout 3 time points.
* The trial will be approved by the institutional view board and conducted in accordance with the principles or Good Clinical Practice guidelines and the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* STAGE CHF BASELINE NYHA functional class II-III and established diagnosis of ischemic cardiomyopathy
* Hospitalization due to acute decompensated CHF
* GDMT for at least 3 months prior to enrollment

Exclusion Criteria:

* Current hospitalization:
* Hemodynamic instability necessitating inotropic or mechanical circulatory support
* Respiratory failure necessitating invasive mechanical ventilation
* Active infection
* A different etiology to explain SIRS other than CHF exacerbation.

Prior hospitalizations or need of intravenous diuretic therapy in the last 30 days before current hospitalization

Cardiac co-morbidities:

Specific HF etiologies:

* Pericardial disease
* Infiltrative myocardial disease
* Moderate and above Valvular heart disease Acute coronary syndrome in the preceding 60 days to randomization Evidence of significant cardiac ischemia within 1 year of randomization without revascularization since Stroke or TIA in the preceding 30 days from randomization

Complex congenital cardiac defect

New initiation of cardiac resynchronization therapy within 60 days prior to randomization

Life threatening arrhythmias /ICD ACTIVATION- in last 90 days Listing for heart transplantation or anticipated/implanted ventricular assist device

Non-cardiac co-morbidities:

* Glomerular filtration rate <30 mL/min/1.73m2 calculated by MDRD formula
* Hepatic insufficiency classified as Child-Pugh B or C
* SBP >180 mm Hg or <110 mm Hg NOT RESPONSIVE TO THERAPY
* Morbid obesity with a BMI >40 kg/m2
* Severe pulmonary disease with requirement of home oxygen therapy or important nocturnal desaturation
* Active treatment for malignancy in the past 2 years or neoplastic spread beyond organ of origin (lymphatic metastases included)
* Hemoglobin <8 g/dL
* Known previous systemic inflammatory disease
* Alcohol or drug abuse Chronic treatment with Copaxone, cytotoxic, immunosuppressant or biological treatment in the past two years.

Known Pregnancy Incapability of signing IC due to cognitive or mental reason Poor compliance to medical therapy or inability to complete the study Age >80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-03-12 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | 3 weeks
  %change in inflammatory cytokines from baseline to Day 3 and 2 weeks (up to 3 weeks), compared between intervention vs. control groups

CONTACTS AND LOCATIONS:
Overall Officials: Offer Amir, PhD, Study Director — Hadassah Medical Centre
Locations (1):
- Hadassah Ein Kerem medical center-hospital ,Cardiology Department, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol